CLINICAL TRIAL: NCT02267499
Title: The Effects of Combined Cognitive and Physical Exercises Through Computer Games in Elderly: The Long Lasting Memories Project (LLM)
Brief Title: Combined Cognitive and Physical Exercises Through Computer Games in Elderly: The LLM Project
Acronym: LLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University of Ulm (Other); Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Assist. Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 84171; 238904 (Other Grant/Funding Number: European Commission Programme CIP-ICTPSP.2008.1.4)
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Healthy
Keywords: cognitive training; physical training; exercise games; novelty serious games; computer training; mild cognitive impairment; mild dementia; healthy elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LLM training (Experimental): Participants use the FitForAll exergaming computer platform as the physical training component (PTC); Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Interventions: Other: LLM training
- Passive Control (No Intervention): Participants do not receive an intervention serving as passive controls

INTERVENTIONS:
Other: LLM training — Participants use the FitForAll exergaming computer platform as the physical training component (PTC); Participants use the language adapted Version of the BrainFitness Program as the cognitive training component (CTC)
  Other Names: PTC+CTC
  Arms: LLM training

SUMMARY:
The study involved Information and Communication Technologies (ICT) and more specifically computer exercises blended with game activities. It was hypothesized that ICT facilitated, game blended combined cognitive and physical exercise improves global cognition when compared to a control group; and that the number of sessions within exercising participants predict cognitive benefits. In addition, we explored the impact of potential moderators on combined exercise-induced cognitive benefits.

DETAILED DESCRIPTION:
The multicenter study was part of the Long Lasting Memories (LLM) project (www.longlastingmemories.eu), which was funded by the European Commission (Information and Communication Technologies Policy Support Program (ICT-PSP) for a three year period (2009-2012). It used a pre-post-test design with the between-participant factor group [intervention vs. passive control]. Post-test was conducted within 2 weeks after completion of the exercise period. Interventions were carried out in Athens and Thessaloniki (Greece) within day care centers, hospitals, senior care centers, a memory outpatient center, local parishes, at university campus facilities (university community installations), and at participants' homes.

Institutions had to provide at least 5 exercise weeks, with a frequency of at least 1 physical and 2 cognitive exercise sessions per week, resulting in at least 5 physical and 10 cognitive exercise sessions in total.

ELIGIBILITY:
Inclusion Criteria:

no severe cognitive impairment [Mini-Mental State Examination, MMSE ≥ 18], fluent language skills, agreement of a medical doctor and time commitment to the test and exercise protocol.

Exclusion Criteria:

concurrent participation in another study, severe physical or psychological disorders which precluded participation in the intervention (i.e., inability to follow instructions), unrecovered neurological disorders such as stroke, traumatic brain injury, unstable medication within the past three months, severe and uncorrectable vision problems, or hearing aid for less than three months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
overall cognition | 2 months
  Greek versions of the California Verbal Learning Test [CVLT], the Digit Span Test and the Trail Making Test [TMT] were used to assess cognitive outcomes.

SECONDARY OUTCOMES:
physical fitness | 2 months
  Physical capacity was measured by means of the Senior Fitness Test
Episodic memory | 2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
working memory | 2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
executive function | 2 months
  calculated by averaging z-standardized sub-scores of the three cognitive tests (primary outcome)
Quality of Life | 2 months
  WHOQoL (WHO Quality of Life)
Instrumental Activities of daily living | 2 months
  IADL
Depressive symptoms | 2 months
  GDS (Geriatric depression scale)
Brain function | 2 months
  changes in abnormal brain waves that correlate with mild cognitive decline and dementia as measured by EEG

REFERENCES:
- See also: The LLM project web site — http://www.longlastingmemories.eu